CLINICAL TRIAL: NCT05288088
Title: Factors Associated With Prolonged In-hospital Stay After Elective Tumor Craniotomy.
Brief Title: Why Still in Neurosurgical Ward After Tumor Craniotomy?
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Alexandra Vassilieva, Medical doctor, PhD-student, Rigshospitalet, Denmark
Other Study IDs: NSwardcraniotomy
Record Dates: First submitted 2022-02-24; First posted 2022-03-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Surgery--Complications; Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Tumor craniotomy patients: Patients undergoing elective brain tumor craniotomy
  Interventions: Diagnostic Test: No intervention

INTERVENTIONS:
Diagnostic Test: No intervention — This is an observational study

SUMMARY:
The aim of this prospective observational study is to identify the specific reasons that prolong a hospital stay after elective tumor craniotomy. Optimal postoperative in-hospital stay is considered to be two days from surgery to discharge from the neurosurgical ward. However, a variable length of stay at a neurological department for follow-up of late recognized deficits of neurological consequences of the surgical procedure are common.

DETAILED DESCRIPTION:
The concept of fast-track surgery and later enhanced recovery after surgery (ERAS) was first imputed in 1990s. Since then, ERAS protocols have been successfully adopted in many surgical fields, often with dramatic benefits for the patients. Length of hospital stay is one of the main questions addressed in many ERAS studies, as it by a simple approach address many of the complications encountered by the patients or the case flow in the perioperative period. Why patients have prolonged hospital stay after surgery has been investigated by Husted et al. in 2011 after hip and knee arthroplasty and P. Munk-Madsen et al. in 2019 after laparoscopic colorectal surgery. Both studies could isolate dominating factors prolonging hospital stay, some of them preventable. Existing length of stay studies on tumor craniotomy patients have focused on specific variables affecting hospital duration, but never explored the true cause of prolonged hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective brain tumor craniotomy

Exclusion Criteria:

* Stereotactic biopsy, pituitary surgery and laser interstitial thermal therapy (LITT)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective tumor craniotomy with the exception of stereotactic biopsy, pituitary surgery and laser interstitial thermal therapy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2022-06-12 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
Hospital length of stay | Patients are followed for a maximum of 6 months.
  Length of stay is defined as the length of inpatient stay, based on number of nights spent at the neurosurgical ward, calculated from the day of surgery to the day of discharge from the neurosurgical ward.

CONTACTS AND LOCATIONS:
Overall Officials: Martin K Sørensen, PhD, Principal Investigator — Department of Neuroanesthesiology, Rigshospitalet
Locations (1):
- Department of Neuroanesthesiology, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided